CLINICAL TRIAL: NCT06370598
Title: A Randomized, Parallel, Open-Label, Phase 1/2a Study to Assess the Safety and Tolerability of Multiple Doses of the Bacteriophage Cocktail TP-122 (Component TP-122A), for the Treatment of Ventilator-Associated Pneumonia
Brief Title: Phase 1/2a to Assess the Safety and Tolerability of TP-122A for the Treatment of Ventilator-Associated Pneumonia
Acronym: RECOVER
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Technophage, SA (Industry)
Collaborators: VectorB2B (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP-122
Record Dates: First submitted 2024-04-10; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Pneumonia, Ventilator-Associated
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TP-122A with SOC (Experimental): Enrolled subjects in the TP-122A+SoC arm will receive IP every 8 hours for 7 days by nebulization and will be followed-up for 28 days after the last IP administration.
  Interventions: Biological: TP-122A
- SOC alone (No Intervention): Just standard of care will be given to patient

INTERVENTIONS:
Biological: TP-122A — Bacteriophage cocktail targeting Psa
  Arms: TP-122A with SOC

SUMMARY:
Given the challenges of treating complex cases of VAP caused by P. aeruginosa and K. pneumoniae, TechnoPhage developed a bacteriophage cocktail (TP-122) against those pathogens, aiming to provide a hospital-based add-on therapy to the SoC including antibiotic therapy, administered by nebulization. TP-122 is a bacteriophage cocktail divided in two different components: TP-122A is comprised of three bacteriophages against infections caused by Pseudomonas aeruginosa and TP-122B includes three bacteriophages against K. pneumoniae . For this study, an effective sample of 15 subjects will be randomly allocated into two arms, in a 3:2 ratio, with 9 subjects receiving TP-122A, in addition to SoC, and 6 subjects receiving the SoC alone.

DETAILED DESCRIPTION:
This is a randomized, parallel, open label, Phase 1/2a study, to assess the safety and tolerability of multiple doses of the component A of the bacteriophage cocktail TP-122 (TP-122A) administered by nebulization in addition to SoC, compared to SoC alone, in adult subjects with VAP. SoC being defined as the treatment dispensed in ICU by the medical team in their usual manner, which will include antibiotic treatment according to current guidelines.

Enrolled subjects randomized to TP-122A arm will receive 5 ml of IP by nebulization, every 8 hours, during 7 days, and will be followed-up for 28 days after the last IP administration.

TP-122 is a bacteriophage cocktail divided in two different components: TP-122A is comprised of three bacteriophages against infections caused by Pseudomonas aeruginosa and TP-122B includes three bacteriophages against K. pneumoniae . B This study will exclusively focus on assessing the safety and effectiveness of component A, TP-122A, specifically targeting infections caused by P. aeruginosa. The IP, TP-122A, will be administered by nebulization at 1x1010 Plaque Forming Units (PFU)/ml every 8h during 7 days, in addition to SoC, for the treatment of adult subjects with VAP due to P. aeruginosa. The decision to go for a frequency of administration of every 8 hours was firstly based on preclinical studies. TP-122A is composed of three lytic bacteriophages targeting P. aeruginosa.

An estimated total of 15 evaluable subjects are expected to complete the study. "Evaluable patients" will be considered subjects that have received at least a total of 9 IP administrations for three consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* 1. Able and willing to sign the ICF. If the subject is unable to do so, the family, a trusted person or a relative should provide consent, as per local regulations.

  2. Subjects with 18 years old, or older.

  3. Subjects with VAP, with stable ventilatory requirements defined as:
* PaO2/FiO2 not lower than 200 mm Hg;
* FiO2 ≤ 0.60
* Compliance not lower than 30 mL/cm H2O;
* Positive End-Expiratory Pressure (PEEP) equal or lower than 10 cm H2O;
* If receiving vasoactive drugs, these must be on a stable dose for the last 24 hours.

AND at least one of the following:

i. Hypoxemia [e.g., PaO2<60 mmHg while the patient is breathing room air, as determined by Arterial Blood Gas (ABG), or worsening of PaO2/FiO2]; and/or ii. Need for acute changes in the ventilator support system to enhance oxygenation, as determined by worsening oxygenation (need to increase FiO2 by 20% or more to maintain oxygen saturation), or needed changes in the amount of PEEP; and/or iii. New onset of suctioned respiratory secretions.

AND at least one of the following signs:

iv. Documented fever (i.e., core body temperature [tympanic, rectal, esophageal] ≥ 38° C [100.4ºF], oral temperature ≥ 37.5°C [99.5ºF], or axillary temperature ≥ 37°C [98.6ºF]); and/or v. Hypothermia (i.e., core body temperature [tympanic, rectal, esophageal] ≤ 35°C [95°F]); and/or vi. White Blood Cell (WBC) count ≥ 10,000 cells/mm³; and/or vii. Leukopenia with total WBC count ≤ 4500 cells/mm³; and/or viii. Greater than 15% immature neutrophils (bands) noted on peripheral blood smear.

4. Microbiological diagnosis of P. aeruginosa infection in the LRT, before randomization.

1. Diagnosis: cultures obtained by Endotracheal Aspirates (ETA), Mini Bronchoalveolar Lavage (BAL) or standard BAL throughout fiberoptic bronchoscopy, subjected to Gram staining and/or Polymerase Chain Reaction (PCR) test (e.g., BIOFIRE® FILMARRAY® Pneumonia Panel plus (Biomerieux)).

   5. Subjects with childbearing potential must have a negative highly sensitive serum pregnancy test at screening.

   Exclusion Criteria:
   * 1. History of any cancer requiring systemic chemotherapy or radiation, in the 5 previous years.

     2. A condition that, in the opinion of the Investigator, could compromise the well-being of the subject, or the course of the study, or prevent the subject from meeting/performing any study requirements/procedures.

     3. Immunocompromised subjects due to illness, organ transplant, or immunosuppressive therapies (e.g., oral or parenteral corticosteroids, methotrexate, immunomodulators), in the last 3 months prior to screening.

     4. Treatment with ad hoc low dose inhaled corticosteroids, in the last 2 weeks prior to randomization (except hydrocortisone and equivalent doses of prednisone and methylprednisolone).

     5. Being pregnant or breastfeeding. 6. Currently participating in another clinical trial or having participated in a clinical trial with receipt of an IP in the last 30 days prior to randomization or in the last '5 half-lives of the IP' prior to randomization (whichever is longer).

     7. Subjects with known community-acquired bacterial pneumonia, or viral or fungal (including Pneumocystis jiroveci) pneumonia (except for subjects that had SARS-CoV-2 related pneumonia more than 6 months before randomization, that do not require Long-Term Oxygen Therapy (LTOT)), or tracheobronchitis (without documented pneumonia), or chemical pneumonitis, or post-obstructive pneumonia (except for subjects with a mild severity disease, that do not require pulmonary function tests); or tracheostomy (except for subjects that have tracheostomy performed while being hospitalised in the ICU).

     8. Subjects requiring Airway Pressure Release Ventilation or High Frequency Oscillatory Ventilation.

     9. Subjects with pleural effusions (or empyema) requiring therapeutic drainage, or lung abscess, or bronchiectasis; or cystic fibrosis, or acute exacerbation of chronic bronchitis, or active pulmonary tuberculosis; or with stage IV congestive heart failure, or cirrhotic liver disease.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate safety and tolerability following nebulization of multiple doses of TP-122A | Day 0, 3 and Day 7
  Analysis of TP-122A arm with SoC versus SoC alone, and individual analysis per treatment arm of the following assessments:
  Adverse Events (AEs):
  1. Incidence of Treatment-Emergent Adverse Events (TEAEs).
  2. Incidence of serious TEAEs. Note: including assessment of seriousness, severity, causality, and outcome.

SECONDARY OUTCOMES:
Proportion of subjects achieving "Clinical Cure" CR | dosing days (1 to 7) and FUp1).
Time to achieve "Clinical Cure" CR | Baseline to EOT
Proportion of subjects achieving "Eradication" or "Presumed Eradication" MR of TP-122A target bacteria | dosing days (1 to 7), FUp1 and FUp2
Time to achieve "Eradication" or "Presumed Eradication" MR | Day o and Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Margarida Barreto, Msc, Study Director — Technophage, SA
Locations (1):
- CH Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided